CLINICAL TRIAL: NCT05442593
Title: The Effect of Biological Maturation on Indices of Exercise-induced Muscle Damage, Neuromuscular Fatigue and Performance After Acute Plyometric Exercise
Brief Title: Biological Maturation and Plyometric Exercise
Acronym: BiMaPlEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Chariklia K. Deli, Assistant Professor, University of Thessaly
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Biol. Matur. - Plyometric Ex.
Record Dates: First submitted 2022-06-23; First posted 2022-07-05 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Biological Maturation
Keywords: children; plyometric exercise; muscle damage; muscle performance; neuromuscular fatigue
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to different groups according to their biological maturation and they will perform the same acute plyometric exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-adolescents (Experimental): Acute plyometric training
  Interventions: Other: Plyometric training
- Adolescents (Experimental): Acute plyometric training
  Interventions: Other: Plyometric training

INTERVENTIONS:
Other: Plyometric training — Participants will perform: 8 sets of 10 maximal countermovement jumps

SUMMARY:
Plyometric training comprises one of the most widely used training methods in both individual and team sports, and is widely used by coaches as one of the main training in both adults, and children. Plyometric training highly includes the component of eccentric contraction. However, eccentric muscle action, especially when unaccustomed, can lead to exercise-induced muscle damage (EIMD), which is accompanied by increased delayed onset of muscle soreness (DOMS), inflammatory responses, increased levels of muscle proteins into the circulation, oxidative stress, and reduction of muscle function and performance the following days. Although plyometric training is widely used in children and may lead to EIMD, there is limited data regarding the acute effects of plyometric exercise training in children. Additionally, the effect of the biological maturation status of children on EIMD after acute plyometric exercise training has not been investigated. The aim of this study is to examine the effect of biological maturation on EIMD after acute plyometric exercise training in children.

DETAILED DESCRIPTION:
Plyometric training comprises one of the most widely used training methods in both individual and team sports. Plyometric training has been shown to improve neuromuscular stimulation, jumping ability, muscle strength, flexibility, muscle mass and muscle performance, running speed and muscle power. Therefore, it is widely used by coaches as one of the main training methods, in both adults, and children).

Plyometric training consists of exercises performed through the stretch-shortening cycle of the muscle where the pre-activated muscle is first stretched (eccentric action) followed by the shortening (concentric) action. Therefore, plyometric training highly includes the component of eccentric contraction. However, eccentric muscle action, especially when unaccustomed, can lead to exercise-induced muscle damage (EIMD). EIMD, amongst others, is accompanied by increased delayed onset of muscle soreness (DOMS), inflammatory responses, oxidative stress, increased levels of muscle proteins and collagen into the circulation, and reduction of muscle function and performance.

The effect of acute plyometric training on EIMD, neuromuscular fatigue and performance has been adequately investigated in adults. Indicatively, an acute protocol of plyometric training increased DOMS, blood inflammatory markers, creatine kinase (CK) and lactate dehydrogenase (LDH) activity, while decreased jumping performance for up to 72 hours after the end of the training. In contrast, data regarding the effect of acute plyometric training on the above indices in children are scarce. Additionally, although some data exist on children versus adults, as far as we know, there is no relative data between children with different stages of biological maturation, regardless the common use of plyometric exercises in youth training. However, such data is crucial for both coaches and young athletes to effectively design the training microcycles and incorporate the training components, but also to reduce the risk of injury.

The aim of the present study is to examine the effect of different biological maturation on EIMD, metabolism, neuromuscular fatigue, oxidative stress, and muscle performance after acute plyometric exercise training in children.

According to a preliminary power analysis (probability error: 0.05, power: 0.80, effect size: 0.30), a total sample of 9 participants per group was considered appropriate in order to detect statistically meaningful changes between groups. Thus, twenty healthy male children, aged 8-15 years old, will participate to the study. Written informed consent will be provided by the parents or legal guardians of children after they will be informed about all risks, discomforts, and benefits involved in the study. The procedures will be in accordance with the 1975 Declaration of Helsinki, as revised in 2013. Approval has been received from the bioethics committee of the Department of Physical Education and Sport Science, University of Thessaly.

The study will be performed in a parallel, repeated measures design. The participants will visit the Department's Exercise Physiology laboratory 9 times in total. During the 1st visit, the participants will be examined by a pediatric endocrinologist in order to estimate their biological maturation and be assigned το a condition of either pre-adolescent or adolescent. A familiarization period with the plyometric training protocol and the evaluation procedures with low intensity will be induced (1st, 2nd, 3rd visit). During the next week (4th and 5th visit), fasting blood samples will be collected in order to estimate testosterone levels, CBC, muscle damage, and oxidative stress markers. Participants will be instructed by a dietitian how to record a 7-days diet recalls to ensure that they do not consume to some greater extent nutrients that may affect EIMD, oxidative stress, and fatigue (e.g. antioxidants, amino acids, etc.). Additionally, assessment of body mass, body height, BMI, body composition, sprint performance, jumping performance, isokinetic strength (concentric, isometric, eccentric), aerobic capacity, EIMD (CK) will be performed. After at least 3 days (6th visit), participants will perform the acute bout of plyometric exercise training, that is 8 sets of 10 maximal squat-jumps with a 2-min rest between sets. DOMS will be estimated prior to and post-training, and lactate concentration prior to, and 4 min after the 4th set and 4 min after the 8th set. Neuromuscular fatigue (maximal voluntary isometric contraction, MVIC) estimation will be performed prior to, and 1 hour, 2 hours, and 3 hours post-training. Additionally, DOMS will be estimated at post-, 24 hours, 48 hours, and 72 hours (7th, 8th, and 9th visit) post-training. Sprint and muscle performance, CBC, CK, and oxidative stress indices will also be estimated at 24 hours, 48 hours, and 72 hours post-training.

ELIGIBILITY:
Inclusion Criteria:

* Normal BMI
* No history of growth irregularities
* No musculoskeletal injuries for at least six months prior to the study
* No use of drugs or ergogenic supplements for at least one month prior to the study
* No participation at exercise with eccentric component for at least three days prior to the study
* No energy drinks consumption before each experimental trial

Exclusion Criteria:

* Abnormal BMI
* History of growth irregularities
* Musculoskeletal injuries in the last six months prior to the study
* Use of drugs or ergogenic supplements in the last month prior to the study
* Participation at exercise with eccentric component in the last three days prior to the study
* Energy drinks consumption before each experimental trial

Ages: 8 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in Creatine kinase | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-plyometric training
  CK will be measured in plasma using a Clinical Chemistry Analyzer with commercially available kits.
Changes in blood lactate | Baseline (pre), 4 minutes post-plyometric training
  Lactate will be measured in capillary blood with a hand-portable analyzer.
Changes in DOMS | Baseline (pre), post-, 24 hours post-, 48 hours post-, 72 hours postplyometric training
  DOMS of knee extensors and knee flexors of both lower extremities will be measured during palpation of the muscle belly and the distal region after performing three repetitions of a full squat and each participant will rate perceived soreness on a scale ranging from 1 (no soreness) to 10 (very sore).
Changes in 10m sprint time | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-plyometric training
  10m sprint time will be measured using light cells Chronojump system
Changes in 30m sprint time | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-plyometric training
  30m sprint time will be measured using light cells Chronojump system
Changes in squat jump | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-plyometric training
  Squat jump height will be measured using a Chronojump contact platform
Changes in counermovement jump | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-plyometric training
  Counermovement jump height will be measured using a Chronojump contact platform
Changes in concentric peak torque | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-plyometric training
  Concentric peak torque of knee extensors and knee flexors will be measured on an isokinetic dynamometer
Changes in eccentric peak torque | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-plyometric training
  Eccentric peak torque of knee extensors and knee flexors will be measured on an isokinetic dynamometer
Changes in isometric peak torque | Baseline (pre), post-, 24 hours post-, 48 hours post-, 72 hours post-plyometric training
  Isometric peak torque of knee extensors and knee flexors will be measured on an isokinetic dynamometer
Changes in maximal voluntary isometric contraction (MVIC) | Baseline (pre), post-, 1 hour post-, 2 hours post-, 3 hours post-plyometric training
  MVIC of knee extensors will be measured on an isokinetic dynamometer

SECONDARY OUTCOMES:
Biological maturation stage | Baseline
  Biological maturation stage will be estimated based on Tanner stage through physical examination by a pediatric endocrinologist
Testosterone levels | Baseline
  Testosterone levels will be estimated via ELISA method with a commercially available kit
Age from Peak Height Velocity (APHV) | Baseline
  APHV will be calculated via an appropriate equation
Body weight | Baseline
  Body weight will be measured on a beam balance with stadiometer
Body height | Baseline
  Body height will be measured on a beam balance with stadiometer
Body mass index (BMI) | Baseline
  BMI will be measured on a beam balance with stadiometer
Maximal oxygen consumption (VO2max) | Baseline
  Maximal oxygen consumption will be estimeted through 20-m shuttle run test
Body fat | Baseline
  Body fat will be measured by using Dual-emission X-ray absorptiometry
Lean body mass | Baseline
  Lean body masswill be measured by using Dual-emission X-ray absorptiometry
Dietary intake | Baseline
  Dietary intake will be assessed using 7-day diet recalls

CONTACTS AND LOCATIONS:
Overall Officials: Chariklia K Deli, PhD, Study Chair — University of Thessaly
Locations (1):
- Department of Physical Education and Sport Science, Uninersity of Thessaly, Trikala, Thessaly, Greece

REFERENCES:
- [Background] Marginson V, Rowlands AV, Gleeson NP, Eston RG. Comparison of the symptoms of exercise-induced muscle damage after an initial and repeated bout of plyometric exercise in men and boys. J Appl Physiol (1985). 2005 Sep;99(3):1174-81. doi: 10.1152/japplphysiol.01193.2004. Epub 2005 Apr 7. PMID 15817716
- [Background] Deli CK, Fatouros IG, Paschalis V, Georgakouli K, Zalavras A, Avloniti A, Koutedakis Y, Jamurtas AZ. A Comparison of Exercise-Induced Muscle Damage Following Maximal Eccentric Contractions in Men and Boys. Pediatr Exerc Sci. 2017 Aug;29(3):316-325. doi: 10.1123/pes.2016-0185. Epub 2017 Feb 6. PMID 28165870
- [Background] Asadi A, Ramirez-Campillo R, Arazi H, Saez de Villarreal E. The effects of maturation on jumping ability and sprint adaptations to plyometric training in youth soccer players. J Sports Sci. 2018 Nov;36(21):2405-2411. doi: 10.1080/02640414.2018.1459151. Epub 2018 Apr 3. PMID 29611771